CLINICAL TRIAL: NCT05109455
Title: Study of a Food Supplement (Mannose and Proanthocyanidins Prolonged Release 24h) Versus Proanthocyanidins in the Prevention of Urinary Tract Infections in Kidney Transplant Patients.
Brief Title: Effects of a Food Supplement in the Prevention of Urinary Tract Infections in Kidney Transplant Patients.
Acronym: MANOTRAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arafarma Group, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ARA-EXP/MN-0801
Record Dates: First submitted 2021-10-21; First posted 2021-11-05 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Kidney Transplant Infection
MeSH Terms: interventions — Dietary Supplements; Proanthocyanidins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food supplement (Experimental): MANOSAR® is an authorized food supplement that contains D-mannose, Proanthocyanidins, Ursolic Acis, vitamin complexes and ions, and protects against urinary tract infections.
  Interventions: Dietary Supplement: MANOSAR®
- Comparator (Active Comparator): The comparator are Proanthocyanidins of continuous-release, which are isolated from cranberry, and prevents the adhesion of uropathogenic bacteria such a E.coli to the wall of the urothelium.
  Interventions: Dietary Supplement: Proanthocyanidins

INTERVENTIONS:
Dietary Supplement: MANOSAR® — MANOSAR® is an authorized food supplement that contains D-mannose, Proanthocyanidins, Ursolic Acis, vitamin complexes and ions, and protects against urinary tract infections.
  Other Names: Food Supplement
  Arms: Food supplement
Dietary Supplement: Proanthocyanidins — The comparator are Proanthocyanidins of continuous-release, which are isolated from cranberry, and prevents the adhesion of uropathogenic bacteria such a E.coli to the wall of the urothelium.
  Arms: Comparator

SUMMARY:
The incidence of Urinary tract infections (UTIs) is very high in kidney transplant patients. Most UTIs occur during the first six months (82% within the first three months) of kidney transplantation and are frequently recurrent. The component D-mannose of our authorized food supplement acts by inhibiting the adherence of E.coli to the urothelium. It also has a controlled release formula that ensures the presence in urine of D-mannose and the other components during 24 hours. This is the reason why this experimental study aims to demonstrate that the oral intake of this food supplement is effective in the prevention of UTIs in kidney transplant patients.

DETAILED DESCRIPTION:
The study tries to analyze the impact of a food supplement (Manosar®) on the incidence of urinary infections in patients undergoing kidney transplantation.

The patients will be randomly distributed (1: 1 ratio) into two treatment groups of 30 patients each. In one group, they will be treated with Manosar®, and in the other group they will be treated with Proanthocyanidins. All patients will be followed for 6 months, being the first three months of the study drug administration.

This experimental study is double-blinded and there are 7 monthly study visits. Properties of D-mannose and Proanthocyanidins make interesting to evaluate the clinical benefit of the use of food supplements with D-mannose and Proanthocyanidins in order to prevent the UTIs without antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years.
* Recipients of a cadaveric donor kidney transplant.
* Patients who are trained to give their informed consent.

Exclusion Criteria:

* Recipients of a kidney transplant who do not authorize their participation in the study by informed consent.
* Recipients of a transplant of an organ other than the kidney.
* Patients with Bricker or Studer neobladders.
* Patients in need of intermittent self-catheterization prior to kidney transplantation.
* Any medical, psychiatric or family condition that, in the opinion of the investigator, may endanger or compromise the patient's ability to participate in the study.
* Pregnant or lactating patients.
* Having participated in clinical trials in the previous 3 months or participating in another clinical study promoted by the pharmaceutical industry, in which the promoter already establishes the treatment for UTI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Change on the incidence of urinary tract infections. | Baseline to 1, 2, 3, 4, 5 and 6 months
  To assess the magnitude of the change from baseline incidence of urinary tract infections in kidney transplant patients at one month, two months and three months of treatment and at four, five and six months of follow-up.

SECONDARY OUTCOMES:
Rate of three types of urinary tract infection: asymptomatic bacteriuria, cystitis, and pyelonephritis between both treatment groups. | Baseline to all study visits up to 6 months.
  All information regarding these infections will be recorded.
Rate of urinary tract infections caused by E.coli. | Baseline to all study visits up to 6 months.
  E. coli will be assessed by urine cultures, which are performed according to the usual clinical practice of the site (weekly - from Visit 0 to Visit 1 (4 urine cultures); fortnightly - from Visit 1 to Visit 3 (4 urine cultures); monthly - from Visit 3 to Visit 6 (3 urine cultures)). Also if there is suspected infection based on clinical criteria there will be performed also an urine culture.
Rate of patients who developed bacteremia during the episode of pyelonephritis. | Baseline to all study visits up to 6 months.
  This will be assessed in relation to the performance of urine cultures.
Rate of safety episodes between both treatment groups. | From Visit 1, and at each visit, up to 6 months.
  All episodes will be recorded, whether considered minor or serious, drug-related or not.
Rate of incidence of delayed renal graft function. | From Visit 0 to Visit 1, up to 1 month.
  This is assessed by the need for a hemodialysis session.
Change from baseline in both treatment groups of concentration of glucose in renal function. | Baseline to all study visits up to 6 months.
  The concentration of glucose (mmol/L) is assessed by the value results of the laboratory analysis, which are completed according to the usual clinical practice of the site for the follow-up of kidney transplant patients: weekly - from Visit 0 to Visit 1 (4 tests); fortnightly - from Visit 1 to Visit 3 (4 tests); monthly - from Visit 3 to Visit 6 (3 tests).
Rate of histologically confirmed acute rejection and number of patients who lost the kidney graft. | Baseline to all study visits up to 6 months.
  Assessed during the 6 months study.
Rate of bacterial colonization of the double J catheter in both treatment groups. | From Visit 0 to Visit 1, up to 1 month.
  This is assessed by the microbiological analysis of the tips of the double J catheter will be performed between Visit 0 and Visit 1, once it has been removed 21-27 days after kidney transplantation.
Type of bacterial colonies of the double J catheter | From Visit 0 to Visit 1, up to 1 month.
  This is assessed by the microbiological analysis of the tips of the double J catheter will be performed between Visit 0 and Visit 1, once it has been removed 21-27 days after kidney transplantation.
Change from baseline in both treatment groups of concentration of Glomerular Filtration Rate (GFR). | Baseline to all study visits up to 6 months.
  The calculation of GFR (ml/min) is estimated with a blood test, which is completed according to the usual clinical practice of the site for the follow-up of kidney transplant patients: weekly - from Visit 0 to Visit 1 (4 tests); fortnightly - from Visit 1 to Visit 3 (4 tests); monthly - from Visit 3 to Visit 6 (3 tests).
Change from baseline in both treatment groups of concentration of serum creatinine in renal function. | Baseline to all study visits up to 6 months.
  The concentration of serum creatinine (µmol/L) is assessed by the value results of the laboratory analysis, which are completed according to the usual clinical practice of the site for the follow-up of kidney transplant patients: weekly - from Visit 0 to Visit 1 (4 tests); fortnightly - from Visit 1 to Visit 3 (4 tests); monthly - from Visit 3 to Visit 6 (3 tests).
Change from baseline in both treatment groups of concentration of sodium in renal function. | Baseline to all study visits up to 6 months.
  The concentration of sodium (mEq/L) is assessed by the value results of the laboratory analysis, which are completed according to the usual clinical practice of the site for the follow-up of kidney transplant patients: weekly - from Visit 0 to Visit 1 (4 tests); fortnightly - from Visit 1 to Visit 3 (4 tests); monthly - from Visit 3 to Visit 6 (3 tests).
Change from baseline in both treatment groups of concentration of potassium in renal function. | Baseline to all study visits up to 6 months.
  The concentration of potassium (mEq/L) is assessed by the value results of the laboratory analysis, which are completed according to the usual clinical practice of the site for the follow-up of kidney transplant patients: weekly - from Visit 0 to Visit 1 (4 tests); fortnightly - from Visit 1 to Visit 3 (4 tests); monthly - from Visit 3 to Visit 6 (3 tests).

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Melilli, Doctor, Principal Investigator — Unidad de Trasplante Renal - Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided